CLINICAL TRIAL: NCT04323618
Title: Investigation of Respiratory-related Tumour Motion in Liver Cancer Patients Undergoing Stereotactic Body Radiotherapy Treatment (SBRT) Using Audiovisual (AV) Biofeedback
Brief Title: Investigation of Respiratory-related Tumour Motion in Liver Cancer Patients Undergoing SBRT Using Audiovisual Biofeedback
Acronym: LAVA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sydney (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: LAVA V4
Record Dates: First submitted 2018-05-03; First posted 2020-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Free breathing or Breathe Well (Other): Free breathing or Breathe Well
  Interventions: Device: Breathe Well

INTERVENTIONS:
Device: Breathe Well

SUMMARY:
Investigation of respiratory-related tumour motion in liver cancer patients undergoing stereotactic body radiotherapy treatment (SBRT) using audiovisual (AV) biofeedback.

ELIGIBILITY:
Inclusion Criteria:

* Liver cancer patients, either primary hepatocellular carcinoma or liver metastases, eligible for stereotactic radiotherapy.
* >18 years old
* Radio-opaque markers implanted (fiducials and/or surgical clips previously implanted in the liver)
* Able to give written informed consent and willingness to participate and comply with the study

Exclusion Criteria:

* Pregnant / lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Improvement in reproducibility of respiratory-related tumour motion (via fiducial maker surrogacy) for liver cancer patients treated with the AV biofeedback respiratory guidance system. | 2 years